CLINICAL TRIAL: NCT07260019
Title: INSTRUMENT ASSISSTED SOFT TISSUE MOBILIZATION VERSUS DRY CUPPING ON UPPER TRAPEZIUS TRIGGER POINTS: A RANDOMIZED CONTROLLED TRIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahim Hassan Elsayed Mohamed Mady, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006052
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Upper Trapezius Trigger Points; Non Specific Chronic Neck Pain
Keywords: IASTM; DRY CUPPING; UPPER TRAPEZIUS TRIGGER POINTS
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study is described as a "single blinded randomized controlled trial". Given the distinct physical nature of the interventions (IASTM vs. Dry Cupping), it is not feasible to blind the participants or the care providers. Blinding will be applied to the Outcomes Assessor, who will perform the outcome measurements without knowledge of the participant's group assignment to prevent bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Control Group) (Active Comparator): Participants will receive a conventional physical therapy program. This includes hot packs applied over the neck and upper shoulders for 15-20 minutes , Transcutaneous Electrical Nerve Stimulation (TENS) applied for 20-30 minutes , and a supervised exercise program (including range of motion, isometric strengthening, chin tucks, and scapular retractions). The treatment will be administered for 3 sessions per week for four weeks.
  Interventions: Other: Hot Packs; Device: Transcutaneous Electrical Nerve Stimulation; Behavioral: Exercise Program
- Group B (IASTM Group) (Experimental): Participants will receive the same conventional physical therapy program as Group A (hot packs, TENS, and exercises) . In addition, they will receive Instrument Assisted Soft Tissue Mobilization (IASTM). This combined treatment will be administered for 3 sessions per week for four weeks.
  Interventions: Device: Instrument Assisted Soft Tissue Mobilization; Other: Hot Packs; Device: Transcutaneous Electrical Nerve Stimulation; Behavioral: Exercise Program
- Group C (Dry Cupping Group) (Experimental): Participants will receive the same conventional physical therapy program as Group A (hot packs, TENS, and exercises) . In addition, they will receive Dry Cupping. This combined treatment will be administered for 3 sessions per week for four weeks.
  Interventions: Device: Dry Cupping; Other: Hot Packs; Device: Transcutaneous Electrical Nerve Stimulation; Behavioral: Exercise Program

INTERVENTIONS:
Device: Instrument Assisted Soft Tissue Mobilization — While the participant is seated, a lubricant (Vaseline) is applied to the skin. The M2T blade is used at a 45° angle to apply slow sweeping strokes along the muscle from origin to insertion (sweeping technique) over the upper trapezius for approximately three minutes.
  Other Names: IASTM , M2T Blade
  Arms: Group B (IASTM Group)
Device: Dry Cupping — While the participant is in a prone position , a single 5cm inner diameter plastic cup is applied to the skin directly over the pre-determined treatment location. The cup is secured by pumping a manual hand-pump three times. The cup is left in place for 5 minutes.
  Arms: Group C (Dry Cupping Group)
Other: Hot Packs — Commercially accessible hot packs (made of bentonite) are placed over the neck and the upper part of the shoulder musculature while the patient is in a prone position. The application lasts for 15-20 minutes.
Device: Transcutaneous Electrical Nerve Stimulation — Applied while the patient is sitting. Electrodes are placed directly over or surrounding the trigger point and along the muscle belly. Parameters: Pulse rate 60-100Hz , Pulse width 40-250 μs. Intensity is set to a tolerable tingling sensation. Treatment duration is 20-30 minutes.
  Other Names: TENS
Behavioral: Exercise Program — A supervised home exercise program consisting of:
  Range of Motion Exercises: Cervical flexion, extension, lateral flexion, rotation, and shoulder shrugs.
  Strengthening Exercises: Isometric cervical flexion, extension, lateral flexion, and rotation; scapular retractions; and chin tucks.
  Dosage: Performed daily for 10-15 repetitions and 2-3 sets

SUMMARY:
The goal of this randomized controlled trial is to compare the effects of Instrument Assisted Soft Tissue Mobilization (IASTM) and dry cupping in patients (both genders), aged 20-50 years, diagnosed with chronic non-specific neck pain who have active upper trapezius trigger points. The main questions it aims to answer are :

1. Is there a significant difference in the effect on pain level (measured by VAS) between the groups?
2. Is there a significant difference in the effect on cervical range of motion (CROM), pressure pain threshold (PPT), and functional disability (NDI) between the groups?

Researchers will compare three groups:

1. Group A (Control):] Will receive a conventional physical therapy program (hot packs, TENS, and exercises).
2. Group B (Experimental):] Will receive conventional therapy plus IASTM.
3. Group C (Experimental):] Will receive conventional therapy plus Dry Cupping.

Participants will be asked to do the following:

1. Undergo baseline assessments (measuring pain, ROM, PPT, and disability) before treatment and final assessments after 4 weeks.
2. Attend [3 treatment sessions per week for four weeks].
3. At each session, all participants will receive the conventional physical therapy program , while Groups B and C will receive their additional intervention (IASTM or dry cupping).

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 20 to 50.
2. Diagnosis of chronic non-specific neck pain (> 4 weeks duration).
3. Had an active upper trapezius TrP (defined as a tender nodule in a taut band that referred pain in a pattern specific for upper trapezius TrP1 or TrP2).
4. Pain of at least 40 mm on a visual analogue scale (VAS).
5. Body mass index from 18 - 30 kg/m2

Exclusion Criteria:

1. Participants who will exhibit signs of fibromyalgia syndrome.
2. Participants with a specific neck pain such as cervical radiculopathy with neurological deficits (e.g., motor weakness, significant sensory loss), cervical instability, fracture, tumor, infection, or inflammatory arthropathies.
3. Sensory problems in the upper or midback regions, heart/circulation problems.
4. Participants who will have vascular syndromes such as vertebrobasilar insufficiency.
5. Participants with skin lesions, fragile skin, or a history of bleeding disorders.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Level | Baseline (before intervention) and after 4 weeks of treatment.
  Pain intensity will be assessed using the Visual Analogue Scale (VAS). The VAS is a self-reported 10 cm line where 0 cm represents "no pain" and 10 cm represents "worst imaginable pain".

SECONDARY OUTCOMES:
Cervical Range of Motion (CROM) | Baseline (before intervention) and after 4 weeks of treatment.
  Active cervical range of motion will be measured in degrees using a Cervical Range of Motion (CROM) device. Measurements will be taken for flexion, extension, lateral flexion (right and left), and rotation (right and left) . Three trials will be averaged for each movement.
Pressure Pain Threshold (PPT) | Baseline (before intervention) and after 4 weeks of treatment.
  PPT will be assessed using a manual pressure algometer applied to the identified myofascial trigger point. Pressure will be increased at a rate of 1 kg/cm² per second until the patient first reports the sensation of pressure changing to pain. The average of three measurements, taken 30 seconds apart, will be recorded.
Functional Disability | Baseline (before intervention) and after the 4-week intervention period.
  Functional disability will be assessed using the validated Arabic version of the Neck Disability Index (NDI-AR). This is a 10-item self-reported questionnaire that evaluates limitations in daily activities and functional impairment due to neck pain.

CONTACTS AND LOCATIONS:
Overall Officials: IBRAHIM H MADY, Bsc, Principal Investigator — Cairo University; Fatma Seddik, Prof.Dr, Study Director — Basic Science Department, Faculty Of Physical Therapy, Cairo University; Ahmed Said, Dr, Study Director — Basic Science Department, Faculty Of Physical Therapy, Cairo University